CLINICAL TRIAL: NCT02832102
Title: Big Data and Models for Personalized Head and Neck Cancer Decision Support (BD2Decide)
Acronym: BD2Decide
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Collaborators: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Amsterdam UMC, location VUmc (Other); Heinrich-Heine University, Duesseldorf (Other); Maastricht Radiation Oncology (Other); Istituto Superiore di Sanità (Other)
Responsible Party: Principal Investigator, Tito Poli, Professor, Azienda Ospedaliero-Universitaria di Parma
Other Study IDs: H2020-PHC30-689715
Record Dates: First submitted 2016-06-01; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Cancer of Head and Neck
Keywords: prognostic modelling; radiomics; clinical decision support system; big data analysis; multiscale prognostic signatures; patient-clinician co-decision tools
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — FFPE tumor specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective cohort: A total of 1000 SCCHN patients will be enrolled in a retrospective observational study treated in the period 2008-2014.
  Standard treatment of SCCHN patients The patients will be managed as foreseen by best clinical practice and international guidelines for SCCHN.
  Interventions: Procedure: Standard treatment of SCCHN patients
- Prospective cohort: A total of 450 SCCHN patients will be enrolled in a study. Each participating Center will select consecutive patients according to the selection criteria (inclusion/exclusion criteria) for one year and will be followed up for two years or more.
  Standard treatment of SCCHN patients: patients will be administered current best clinical practice treatments.
  Interventions: Procedure: Standard treatment of SCCHN patients

INTERVENTIONS:
Procedure: Standard treatment of SCCHN patients — The interventions may include surgery, radiotherapy, chemotherapy or combined therapies, as recommended by best practice and international guidelines.

SUMMARY:
The purpose of this study is to determine new multiscale signatures for the prediction of head and neck cancer (HNC) patients disease outcome, in particular for advanced stage (stage III, IV) human papillomavirus (HPV) negative patients and to validate prognostic models for overall survival.

DETAILED DESCRIPTION:
The clinical study is devoted to the validation of a decision support system for HNC patients management in the frame of a H2020 project.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Histologically confirmed diagnosis of oral cavity, oropharynx, larynx, hypopharynx squamous cell carcinoma
* Clinical stage III and IV
* Patient candidate for curative treatment: ± surgery ± radiotherapy ± chemotherapy
* Adequate archival pre-treatment tumor specimen available (FFPE macrodissected sections)
* Availability of baseline diffusion-weighted imaging (DWI) - Magnetic Resonance Imaging (MRI) acquisition (non-TRACE ) with more than 3 b-values (ranging from 0 (included) to 1000 s/mm2), and a field map acquisition.
* MRI images, T1 and T2 weighted, (slice thickness lower than 3 mm), head and neck in a single volume, and/or CT scan of the head and neck performed with contiguous cuts of 2-3 mm or less in slice thickness with i.v. contrast
* Male or female ≥ 18 years old

Exclusion Criteria:

* Any previous haed and neck cancer.
* Patients with previous malignancies in the last 5 years before treatment for head and neck cancer, with the exception of surgically cured carcinoma in situ of the cervix, in situ breast cancer, incidental finding of stage T1a or T1b prostate cancer, and basal/squamous cell carcinoma of the skin.
* Any previous malignancy that was treated with surgery and or radiation of the head and neck region.
* Histological type other than head and neck squamous cell cancer (nasopharynx, salivary glands and sinus nasal cancer are excluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective study cohort: A total of 450 SCCHN patients Stage III and IV, followed up for 18-24 months or more.
  Retrospective study cohort: A total of 1000 SCCHN patients Stage III and IV, diagnosed between year 2008 and 2014.
Sampling Method: Non-Probability Sample
Enrollment: 1450 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Realizes and validates an Integrated Decision Support System (BD2Decide platform) | through study completion, an average of 3 year
  The primary endpoint of this study is the accuracy of the prediction of prognosis based on the BD2Decide platform compared to Tumor Node Metastasis staging (in a population consisting of patients with different subtypes of head and neck cancer).

SECONDARY OUTCOMES:
Improved Quality of Life | baseline, month 6, month 18, month 24 after primary treatment
  To measure patients' QoL in relation to the new prognostic stratification
Assess survival time | at 2, 3 and 5 years
  Overall survival and disease free survival will be assessed to verify the accuracy of the prediction of BD2Decide platform

CONTACTS AND LOCATIONS:
Overall Officials: Tito Poli, MD, PHD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma
Locations (5):
- Heinrich-Heine Universitaet Dusseldorf, Dept. of Othorinolaryngology, HHU, Düsseldorf, Germany
- Italy (2):
  - Fondazione Irccs Istituto Dei Tumori Milano, Milan, MI
  - Azienda Ospedaliero Universitaria di Parma, Parma, PR
- Netherlands (2):
  - Stichting VU/VUmc, Amsterdam
  - Maastricht Radiation Oncology MAASTRO Clinic, Maastricht

IPD SHARING:
Plan to Share IPD: Yes
Patients' data are pseudonymised and stored in a shared Case Report Form (CRF) for data analysis

REFERENCES:
- [Derived] Cavalieri S, Brakenhoff RH, Leemans CR, Hoebers FJP, Poli T, Scheckenbach K, Iacovelli NA, Franceschini M, Orlandi E, Licitra L, De Cecco L. Prognostic gene expression signatures for HPV-negative head and neck squamous cell carcinoma. Radiother Oncol. 2025 Jul;208:110900. doi: 10.1016/j.radonc.2025.110900. Epub 2025 Apr 17. PMID 40252811
- [Derived] Cavalieri S, Serafini MS, Carenzo A, Canevari S, Brakenhoff RH, Leemans CR, Nauta IH, Hoebers F, van den Hout MFCM, Scheckenbach K, Hoffmann TK, Ardighieri L, Poli T, Quattrone P, Locati LD, Licitra L, De Cecco L. Clinical Validity of a Prognostic Gene Expression Cluster-Based Model in Human Papillomavirus-Positive Oropharyngeal Carcinoma. JCO Precis Oncol. 2021 Oct 27;5:PO.21.00094. doi: 10.1200/PO.21.00094. eCollection 2021. PMID 34738049